CLINICAL TRIAL: NCT02967198
Title: Pre-procedure Planning for Liver Biopsy or Radiofrequency Ablation Using the Automatic Fusion Images of the Registrated 3D CT or MR-US Scans
Brief Title: Pre-procedure Planning for Liver Biopsy or Radiofrequency Ablation Using CT or MR/US Fusing Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508-099-695
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Liver Mass; Liver Fibroses
Keywords: Fusion; Ablation; Percutaneous biopsy; Shear wave elastography
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT/US fusion (Experimental): patients undergo routine conventional feasibility planning ultrasound, and clinical decision of percutaneous liver biopsy or RFA feasibility is made based on conventional planning ultrasound. Then additional planning ultrasound using CT/US fusion technique is immediately performed by the same operator, and clinical decision is made based on fusion imaging.
  Interventions: Device: CT/US fusion; Device: ultrasound shear wave elastography

INTERVENTIONS:
Device: CT/US fusion — Fusion of pre-procedure cross-sectional imaging (CT or MRI) and real-time USG using registration function of USG device.
Device: ultrasound shear wave elastography — ultrasound shear wave elastography is performed in S-shear wave scanner according to guidelines of ultrasound elastography.
  Other Names: S-shear wave

SUMMARY:
The purpose of this study is to determine whether fusion technique of preradiofrequency ablation (RFA) or percutaneous liver biopsy cross-sectional imaging (CT or MR) and real-time ultrasonography would improve feasibility of RFA or liver biopsy in patients with liver tumor in comparison with ultrasonography guidance alone. And assessment of a new point shear-wave elastography method (pSWE, S-shear wave) and compare its accuracy in assessing liver stiffness (LS) with another pSWE technique (ARFI).

DETAILED DESCRIPTION:
RFA is one of commonly used local therapies for primary or secondary liver tumors. And percutaneous liver biopsy is very important technique to confirm the diagnosis of focal hepatic lesion whether benign or malignancy.

For successful and safe procedure, safe access route and lesion visibility are essential , and the conditions are usually evaluated on pre-procedure planning ultrasonography (USG). However, these procedure is sometimes aborted due to limited sonic window of various cause and challenging identification of small isoechoic tumors or hepatocellular carcinomas among dysplastic nodules . Therefore, precise targeting and assuring safe route would be of clinical importance. In this preliminary study, investigators attempted to determine US and CT/MR fusion technique would be able to improve RFA or liver biopsy feasibility in patients with liver tumors in comparison with conventional US alone technique.

In addition, to assess intra- and inter-observer reproducibility of a new point shear-wave elastography method (pSWE, S-shear wave) and compare its accuracy in assessing liver stiffness (LS) with another pSWE technique (ARFI).

ELIGIBILITY:
Inclusion Criteria:

* all conditions should be satisfied for inclusion.

  * referred to Radiology in our institution for liver tumor RFA or percutaneous liver biopsy
  * available pre-procedure liver CT or liver MR imaging within 6 weeks

Exclusion Criteria:

* any contraindication of liver RFA or percutaneous liver biopsy • any patients who received treatment between pre-RFA imaging and planned RFA.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
RFA or biopsy feasibility rates on planning USG with/without fusion CT/MR and US | 10 minutes after finishing planning USG
  comparison of rates of RFA feasibility on conventional planning USG and on fusion planning USG
Assessment of a new point shear-wave elastography method (pSWE, S-shear wave) | 10 minutes after finishing planning USG
  To assess intra- and inter-observer reproducibility of a new point shear-wave elastography method (pSWE, S-shear wave) and compare its accuracy in assessing liver stiffness (LS) with another pSWE technique (ARFI).

SECONDARY OUTCOMES:
Rate of tumor visibility on planning USG with/without fusion technique | 10 minutes after finishing planning USG
  comparison of tumor visibility (or detection) rates on planning USG on conventional planning USG and fusion planning USG
Number of patients with safety access route on planning USG with/without fusion technique | 10 minutes after finishing planning USG
  comparison of number of patients with presence/absence of safety access route, and the on two planning USGs

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No